CLINICAL TRIAL: NCT05293925
Title: Consultation d'Annonce d'Arrêt de la Chimiothérapie et Des Traitements Spécifiques en Contexte Ambulatoire: évaluation de l'Impact Psychologique et Des échanges d'Informations.
Brief Title: Consultation to Announce the End of Chemotherapy and Specific Treatments in an Outpatient Setting: Evaluation of the Psychological Impact and Information Exchange.
Acronym: CACTuS
Status: Completed | Type: Observational
Sponsor: Institut Curie (Other)
Responsible Party: Sponsor
Other Study IDs: IC2021-14
Record Dates: First submitted 2022-02-25; First posted 2022-03-24 (Actual); Last update posted 2023-12-19 (Actual); Status verified 2023-12

CONDITIONS: Cancer
Keywords: Quality of end of life; Palliative care; Announcement of cessation of treatment
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: announcement of cessation of treatment — The first 40 outpatients for whom an announcement to stop anti-tumour treatments is made at the Institut Curie Paris, in a conventional oncology consultation or in Palliative Care Day Hospital.
  Categorical variables will be described by numbers and percentages. Quantitative variables will be described by the mean, standard deviation, median of the distribution as well as the minimum, maximum and interquartile range and compared by a Student's t test or a Wilcoxon test according to the normality of the variables.

SUMMARY:
The average 5-year survival rate for patients diagnosed with cancer in France is estimated at 53%. Nearly half of all patients diagnosed with cancer are not alive 5 years after diagnosis Discontinuation of anti-tumor treatments is therefore a major issue in their care. Discussing the discontinuation of specific treatments requires scientific oncological skills but also communication skills. The difficulties encountered by oncologists concerning communication about the end of life are linked to the doctors' personal discomfort with death, their fear of the responsibility of stopping chemotherapy, and their distrust of their colleagues. On the other hand, they may also come from patients who are supposedly reluctant to talk about the end of life, a reluctance that is heightened in the case of language barriers, young age or pressure from families. Finally, the place of practice could explain some of the difficulties in talking about the end of life, notably because of a lack of training in delivering bad news or a stigma attached to palliative care.

This exploratory work should make it possible to describe the characteristics of the announcement of the cessation of anti-tumor treatments in ambulatory patients, to evaluate distress, anxiety, depressive symptomatology, as well as the satisfaction of the patients concerning the management received.

DETAILED DESCRIPTION:
In this pilot study, we will describe for the first time the discontinuation of anti-tumour treatments in outpatients with advanced cancer and evaluate the psychological impact on patients following this announcement.

In outpatients patients, these announcements of treatment cessation will be made in a conventional oncology consultation or in Palliative Care Day Hospital.

This exploratory work should make it possible to describe the characteristics of the announcement of the cessation of anti-tumour treatments in ambulatory patients, to assess distress, anxiety, and the depressive symptomatology, as well as patient satisfaction with the treatment received.

The 2 hypotheses of this research work are the following:

1. the announcement of the cessation of specific treatments can generate distress, anxiety and depressive symptoms for the patient, and may be a source of dissatisfaction with the quality of care received.
2. the existence of an improvement in the quality of the announcement when it is made in HDJ SP in comparison with an announcement made in a conventional oncology consultation; reduction of the psychological impact for the patient, reduction in markers of aggressiveness of care at the end of end of life care. The doctors involved in this project have received training in listening to and supporting patients with advanced cancer in a palliative situation.

ELIGIBILITY:
Inclusion Criteria:

* Major outpatients with advanced cancer for whom anti-tumour treatment is announced by the oncologist in a conventional oncology consultation or in Palliative Care Day Hospital.
* Patient who speaks and understands the French language.
* Patient over 18 years of age.
* Patient informed and not opposed.

Exclusion Criteria:

* Refusal of the patient or doctor to participate in the study.
* Patient does not speak or understand the French language.
* Patient under 18 years of age.
* Persons deprived of liberty or under guardianship (including curatorship).
* Persons of legal age under court protection.
* Inability to participate in the study for geographical, social or psychological psychological reasons.

Ages: 18 Years to 125 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chronological inclusion of the first 40 outpatients for whom an announcement to stop anti-tumour treatments was made at the Institut Curie Paris, in a conventional oncology consultation or in a Palliative Care Day Hospital
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2022-01-27 (Actual); Primary Completion 2023-07-25 (Actual); Study Completion 2023-07-25 (Actual)

PRIMARY OUTCOMES:
Emotions thermometers | Baseline
  It will be offered to the patient before and after the announcement of the cessation of treatment, as well as on the 7th day after the announcement of the end of anti-tumour treatments.These thermometers have a scale of 0 to 10 and will indicate the average level of distress, anxiety, depression, anger, and help needed for the past week including the current day. Higher scores mean a worse outcome
Emotions thermometers | Day 0
  These thermometers have a scale of 0 to 10 and will indicate the average level of distress, anxiety, depression, anger, and help needed for the past week including the current day. Higher scores mean a worse outcome
Emotions thermometers | Day 7
  These thermometers have a scale of 0 to 10 and will indicate the average level of distress, anxiety, depression, anger, and help needed for the past week including the current day. Higher scores mean a worse outcome

SECONDARY OUTCOMES:
Hospital Anxiety and Depression Scale (HADS) | Baseline
  The HAD is a 14-item questionnaire, with two 7-item subscales, assessing anxiety and depression respectively. Each item is scored from 0 to 3, for a total score of 21 per subscale and 42 for the total HADS. Thus a high total score correlates with a high intensity of anxiety and depression
Hospital Anxiety and Depression Scale (HADS) | Day 7
  The HAD is a 14-item questionnaire, with two 7-item subscales, assessing anxiety and depression respectively. Each item is scored from 0 to 3, for a total score of 21 per subscale and 42 for the total HADS. Thus a high total score correlates with a high intensity of anxiety and depression
EORTC QLQ PATSAT-C33 (Questions 1 to 10) | Day 7
  This questionnaire explores the area of care provided by physicians. The doctor section comprises three sub-domains addressing technical skills (3 items), information exchange (3 items), and affective behaviour (4 items). Each item is scored from 1 to 5. Higher scores mean a better outcome

CONTACTS AND LOCATIONS:
Overall Officials: Romain SEBAN, MD, Principal Investigator — Instiut Curie
Locations (1):
- Institut Curie, Paris, France